CLINICAL TRIAL: NCT04596514
Title: A Randomised Trial on Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-traumatic Out of Hospital Cardiac Arrest
Brief Title: Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-traumatic Out of Hospital Cardiac Arrest
Acronym: REBOARREST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1253-0322; U1111-1253-0322 (Registry Identifier: WHO Universal Trial Number UTN)
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest
Keywords: Reboa procedure; aortic occlusion; resuscitation; pre-hospital emergency care
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded from the statisticians who carry out analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - REBOA (Experimental): Resuscitative Balloon Occlusion of the Aorta after advanced cardiac life support if return of spontaneous circulation is not achieved
  Interventions: Procedure: REBOA; Procedure: usual procedure according to guidelines
- Control group - ACLS (Active Comparator): Advanced cardiovascular life support as described in the guidelines
  Interventions: Procedure: usual procedure according to guidelines

INTERVENTIONS:
Procedure: REBOA — Resuscitative endovascular balloon occlusion of the aorta (REBOA)
  Arms: Intervention group - REBOA
Procedure: usual procedure according to guidelines — Treatment as described in the guidelines from the European Resuscitation Council, the Norwegian Resuscitation Council, and other local national guidelines

SUMMARY:
The primary aim of this trial is to assess the efficacy of resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct treatment to advanced cardiovascular life support (ACLS) in patients with out-of-hospital cardiac arrest.

Out of hospital cardiac arrest (OHCA) carries a high mortality rate. The treatment of out-of-hospital cardiac arrest is ACLS as stated in the guidelines from the Norwegian Resuscitation Council and the European Resuscitation Guidelines.

Recently, REBOA has been proposed as an adjunct treatment in management of non-traumatic cardiac arrest patients, because thoracic aortic occlusion provides a redistribution of the cardiac output to organs proximal to the occlusion. Preclinical studies demonstrate that REBOA during CPR provide both increased coronary artery blood flow and perfusion pressure and increased rates of return of spontaneous circulation (ROSC).

This is the first prospective trial in the world to assess the efficacy of REBOA in non-traumatic cardiac arrest. The intervention is shown feasible in the pre-hospital setting. If this trial provides a signal of benefit in patients, this study could initiate further clinical research which could change current resuscitation practice world-wide.

DETAILED DESCRIPTION:
This is a prospective, randomised, parallel group, multi-centre, phase II clinical trial.

Patients are randomised in a 1:1 ratio to be included to the control group or the intervention group. The control group receives ACLS according to national guidelines, while the intervention group receives ACLS according to national guidelines and the REBOA procedure as an adjunct treatment.

The REBOA procedure is performed by a team consisting of a physician (anesteshiologist) and a paramedic, working at a helicopter emergency medical service (HEMS) base. All operators will be properly educated and tested before they can include patients.

If the patients in the intervention group achieves ROSC, the balloon will be deflated and post-ROSC treatment will be continued as per routine.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest
* non-traumatic cardiac arrest
* less than 10 minutes from debut of arrest to start of basic or advanced cardiac life support
* advanced cardiac life support is established and can be continued

Exclusion Criteria:

* traumatic cardiac arrest, including strangulation, electrocution and patients rescued from avalanches
* accidental hypothermia with temperature < 32 0C
* suspected cerebral hemorrhage as etiology of the arrest
* suspected non-traumatic hemorrhage as etiology of the arrest
* pregnancy, obvious or suspected
* patient included to the study site's E-CPR protocol
* other factors as decided by the treatment team (environmental factors, safety factors and others)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that achieve return of spontaneous circulation (ROSC) with a duration of at least 20 minutes. | 60 minutes
  Sustained ROSC means return of spontaneous circulation with a duration of at least 20 minutes.

SECONDARY OUTCOMES:
The proportion of patients surviving to 30 days with good neurologic status, defined as a modified Rankin scale (mRS) score 0-3. | 30 days
  The mRs are dichotomised into good (score 0-3) and poor (score 4-6) neurological state.
Difference in end-tidal CO2 (EtCO2) measurements between control group and intervention group after aortic occlusion. | 15 minutes
  In the control group, EtCO2 is measured after airway management is completed. In the intervention group, EtCO2 is measured after airway management is completed, before balloon inflation and 30, 60 and 90 seconds after balloon inflation.
Change in blood pressures after aortic occlusion | 15 minutes
  In the intervention group, intra-aortic blood pressure measurements from the REBOA catheter are recorded. This applies only to the catheters with CE/FDA approval for invasive blood pressure measurements and will therefore be assessed in a sub-group of the participants. Continuous registration of invasive blood pressure will start before aortic occlusion.
Difference in left ventricular ejection fraction (LVEF) measured by echocardiography | 1-2 weeks
  Echocardiography after admission, after a few days-up to one week and at discharge will be assessed - both from the control and intervention group.

OTHER OUTCOMES:
Exploratory outcome - All-cause mortality one year after randomization | One year
  Difference in all-cause mortality between the intervention and control group after one year.
Exploratory outcome - Difference in renal function between intervention and control group | 30 days
  Values of serum creatinine (umol/L) and urine output (ml/kg/h) will be combined to classify renal function according to the Acute Kidney Injury Network (AKIN) classification, into stage 1-3.
Exploratory outcome - difference in the need for renal replacement therapy between intervention and control group | 30 days
  Number of days renal replacement therapy is needed
Exploratory outcome - difference in the liver function (albumine) between intervention and control group | 30 days
  Value of albumine (mg/L)
Exploratory outcome - difference in the liver function (ASAT/ALAT) between intervention and control group | 30 days
  Value of ASAT and ALAT (U/L)
Exploratory outcome - Incidents of all adverse events | 30 days
  assessment of all adverse events, both suspected and unsuspected, in both intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, MD, PhD, Study Director — St Olav's Hospital
Locations (11):
- Denmark (4):
  - Aarhus Base, Aarhus
  - Billund HEMS-base, Billund
  - Ringsted HEMS-base, Ringsted
  - Skive HEMS, Skive
- Maggiore Hospital, Bologna, Italy
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Drammen Hospital, Drammen
  - Lørenskog HEMS Unit, Oslo
  - Rapid response car - 119 Oslo, Oslo
  - Stavanger University Hospital, Stavanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol, statistical analysis plan, information letter for consent and other trial documents will be published open access. The clinical study report and statistical analysis report will also be made openly available but may be altered to hide information that may lead to identification of individual study participants. These documents will be shared at HUNT Cloud.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and ICF will be available before study start. SAP will be available before first interim analysis.
Access Criteria: Individual level data will be made available to sponsor institutions on the REBOARREST data space in HUNT Cloud. Access will be controlled by a data processor agreement between the partner and funder. Pseudonymous individual level data collected during the trial, will be made available on request to researchers from other scientific institutions by approval of the project management to ensure that usage is compliant with privacy and consent requirements as well as conditions for attribution and usage.
  Data sharing with editors or peer-reviewers of scientific journals, conferences or the like will not require additional consent or data access agreement with sponsor, as such data will not be shared onward or used beyond reviewing this trial.
  After data sharing, the sponsor must be acknowledged in any publication resulting from the shared data. For closer collaboration attribution based on the Vancouver Convention will apply.
URL: http://www.reboarrest.com

REFERENCES:
- [Background] Brede JR, Lafrenz T, Klepstad P, Skjaerseth EA, Nordseth T, Sovik E, Kruger AJ. Feasibility of Pre-Hospital Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2019 Nov 19;8(22):e014394. doi: 10.1161/JAHA.119.014394. Epub 2019 Nov 11. PMID 31707942
- [Derived] Brede JR, Skulberg AK, Rehn M, Thorsen K, Klepstad P, Tylleskar I, Farbu B, Dale J, Nordseth T, Wiseth R, Kruger AJ. REBOARREST, resuscitative endovascular balloon occlusion of the aorta in non-traumatic out-of-hospital cardiac arrest: a study protocol for a randomised, parallel group, clinical multicentre trial. Trials. 2021 Jul 31;22(1):511. doi: 10.1186/s13063-021-05477-1. PMID 34332617